CLINICAL TRIAL: NCT03778515
Title: Novel Quantitative MRI for Axial Spondyloarthritis
Status: Terminated | Type: Observational
Why Stopped: Lack of enrollment due to the pandemic
Sponsor: The Cleveland Clinic (Other)
Collaborators: University of California, San Francisco (Other); UCB PHARMA Inc. (US) (Industry)
Responsible Party: Principal Investigator, Xiaojuan Li, Xiaojuan Li, PhD, Professor, Department of Biomedical Engineering, The Cleveland Clinic
Other Study IDs: 18-1327
Record Dates: First submitted 2018-11-27; First posted 2018-12-19 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Spondylitis, Ankylosing
Keywords: Axial; Spondyloarthritis; MRI; Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing; Spondylarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cases - Ankylosing Spondylitis Cohort: 20 patients with ankylosing spondylitis (AS). Fifteen of these patients will be recruited from the Ankylosing Spondylitis clinic at the University of California, San Francisco. Five patients will be recruited from the Rheumatology clinic at the Cleveland Clinic. Observational with MRI.
  Interventions: Diagnostic Test: MRI
- Controls - w/o Ankylosing Spondylitis: 5 patients without AS and with no history of any arthritis or lower back pain in this study. These 5 patients will make up the control group of the study, which means that they will provide a benchmark of comparison for the results investigators obtain from the active AS group. 2 of these 5 patients will be recruited from Cleveland Clinic, and 3 will be recruited from UCSF. Observational with MRI
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Observational Study of novel MR imaging and image processing techniques that will provide reliable and fully quantitative evaluation of inflammation, chronic structural changes and vascularity in patients with Ankylosing Spondylitis (AS).

SUMMARY:
This proposal aims to develop novel MR imaging and image processing techniques that will provide reliable and fully quantitative evaluation of inflammation, chronic structural changes and vascularity in patients with Ankylosing Spondylitis (AS). The quantitative evaluation will be more objective and reproducible, more sensitive to subtle changes, and less time consuming, as compared to the current semi-quantitative evaluation. It will allow radiologists and rheumatologists to evaluate the inflammation and structural changes more reliably to improve early diagnosis and treatment response evaluation. The developed quantification tools can be disseminated to other research and clinical sites for retrospective and prospective data analysis, and used as outcome measures for future multi-center trials. The evaluation of vascularity will enhance Investigators understanding of disease pathophysiology and serve as a novel marker to improve investigators capability of evaluating and predicting treatment response in AS. The successful implementation will greatly assist clinicians to optimize individualized therapeutic strategies and ultimately improve patient care for AS.

DETAILED DESCRIPTION:
There is a critical and unmet clinical need for non-invasive techniques that provide early diagnosis as well as reliable and sensitive evaluations of ongoing disease activity and treatment response in patients with axial spondyloarthritis (axSpA). Imaging plays a key role to fulfill this goal and there is an increasing trend of applying imaging techniques in the field of axSpA. However, current imaging techniques, including radiographs and MRI, are primarily limited to qualitative or semi-quantitative evaluations of disease activity and structural damage, which is very crude and subjective with considerable inter-reader variation, and has limited sensitivity of detecting early lesions as well as changes in inflammatory lesions beyond morphology of bone marrow edema after treatment. Furthermore, several recent studies reported data of inflammation (bone marrow edema), fatty deposition and new bone formation after TNF inhibitor (TNFi) treatment in patients with axSpA, suggesting a complex relationship between inflammation, bone formation, and suppression of the TNF pathway. These studies also call for differentiating edema for their characteristics (angiogenesis for example) and inflammation stages (acute and chronic), which will provide valuable insight on disease pathophysiology as well as on optimizing treatment for individual patients with axSpA.

The long-term goal is to develop novel quantitative MRI measures that will reliably assess both inflammation and structural damage, and predict treatment response, remission and disease progression in axSpA. Compared to current MRI grading systems, such quantitative measures may be used as more sensitive, specific, reliable and faster imaging markers for future trials, and eventually for clinical practice to improve patient management in axSpA. In this proposal, Investigators will focus on patients with clinically diagnosed active Ankylosing Spondylitis (AS) and will develop novel imaging and image processing techniques using 3 Tesla MRI. The specific aims are two-folds. Firstly, Investigators will develop methods that reliably quantify bone marrow edema (BME), fatty deposition (FD) and erosions; Secondly, Investigators will develop novel quantitative evaluation of perfusion and vascularity of BME (using dynamic Gd-enhanced MRI), which has not been investigated for axSpA in the literature.

Investigators will recruit 20 patients with active Ankylosing Spondylitis (AS) using the 1984 modified NY criteria. Fifteen patients will be recruited from the Ankylosing Spondylitis clinic at UCSF, directed by Dr. Lianne Gensler, and five patients will be recruited from Rheumatology clinic at the Cleveland Clinic by Dr. Elaine Husni. Drs. Gensler and Husni will also reach out to the other academic sites and the community private practices to recruit patients as needed who are starting TNF inhibitor therapy with CZP for their AS. Patients will be studied at baseline, 4-weeks and 48-weeks after initiation of TNFi treatment. Advanced quantitative MRI will be applied to evaluate early treatment response at 4-weeks, and long-term outcomes at 48-weeks. The central hypothesis is that quantitative MRI allows a fast, specific and reproducible evaluation of disease activity and structural changes in AS, and provides more superior diagnostic and prognostic capability compared to semi-quantitative MRI grading systems.

The successful implementation of the proposed study will make significant contributions to the research and clinical

ELIGIBILITY:
Inclusion Criteria:

* Active AS meeting the modified New York criteria
* BASDAI ≥ 4
* Elevated C-Reactive Protein
* ≥ 18 years old
* Initiation of TNFi treatment with CZP

Exclusion Criteria:

* Previous treatment with more than one biologics
* Biologic treatment within six-months (no more than 20% of group (n=4) for patients with previous biologic treatment)
* Non-response to previous anti TNF treatment
* Fibromyalgia or other reasons for back pain
* Pregnant patients
* Patients on > 10mg of Prednisone per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 15 patients will be recruited from the Ankylosing Spondylitis clinic at UCSF, and five patients will be recruited from Rheumatology clinic at the Cleveland Clinic. 10 patients with disease duration <= 10 years, and ten patients with disease duration > 10 years but without complete ankylosis. 5 healthy controls will be recruited for evaluating the measurement, with 2 from CCF and 3 from UCSF. The volunteers will be studied at baseline and 1-year follow up.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Volume of MRI bone marrow edema (in cm^3) from Baseline at 48-weeks | Change from Baseline at 48-weeks
  Fully quantitative evaluation of volume of bone marrow edema (in cm^3) will be developed and applied in the study. Volume of BME will be calculated in both SIJ and Spine in high-resolution MR images to evaluate the active inflammation in the patients.
Change in MRI grading SPARCC from Baseline at 48-weeks | Change from Baseline at 48-weeks
  Inflammation and structural damages, including bone marrow edema, fatty deposition, erosions, syndesmophytes and ankylosis, in the spine and SIJs will be graded in MR images by certified radiologists using validated scoring systems developed by the Spondyloarthritis Research Consortium of Canada (SPARCC).

SECONDARY OUTCOMES:
Change in C-reactive protein (CRP) (in mg/dL) from Baseline at 48-weeks | Change from Baseline at 48-weeks
  CRP will be measured for evaluating inflammation activity.
Change in Ankylosing Spondylitis Disease Activity Score (ASDAS)-CRP at Baseline, 4-weeks, 48-weeks | Change from Baseline at 48-weeks
  The Ankylosing Spondylitis Disease Activity Score (ASDAS) is a new composite index to assess disease activity in Ankylosing Spondylitis (AS). It combines five disease activity variables with only partial overlap, resulting in one single score with better truth (validity), enhanced discriminative capacity and improved sensitivity to change as compared to single-item variables. ASDAS-CRP will be calculated as 0.12 x Back Pain + 0.06 x Duration of Morning Stiffness + 0.11 x Patient Global + 0.07 x Peripheral Pain/Swelling + 0.58 x Ln(CRP+1).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojuan Li, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- University of California, San Francisco, San Francisco, California, United States